CLINICAL TRIAL: NCT03355703
Title: Results of Anterior Odontoid Screw Osteosynthesis in Treatment of Type 2 Odontoid Fracture
Brief Title: Anterior Odontoid Screw Osteosynthesis in Treatment of Type 2 Odontoid Fracture
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed mohamed fayez, Principal investigator Ahmed mohamed fayez, Assiut University
Other Study IDs: Trauma unit
Record Dates: First submitted 2017-10-21; First posted 2017-11-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Odontoid Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Odontoid fracture is a common fracture accounting for 10-15% of all cervical fractures. It occurs in bimodal fashion in elderly and young patients.

The classification of Anderson and Alonzo provides a guide for prognosis . Type I and type III have a good rate of union, while type II has a poor prognosis due to poor blood supply. Hence, operative fixation is recommended to avoid non-union.

Treatment options for type II include anterior odontoid screw fixation and posterior C1-C2 fusion.Despite the excellent rates of bony union in posterior C1-C2 fusion, it is associated with higher morbidity, higher blood loss and significant limitation in the range of motion and rotation of the neck.the aim of the study Is to evaluate clinical and radiological outcome of anterior odontoid screw osteosynthesis in treatment of type 2 odontoid fracture.

DETAILED DESCRIPTION:
Preoperative evaluation:

Full clinical Evaluation and management in trauma unit using Advanced Trauma Life Support protocols.

Full neurological assessment and classification using American Spinal Injury Association score.

Radiological assessment includes antero-posterior and lateral plain cervical radiograph and CT scan for all patients. MRI will be done neurological deficit

Operative technique:

Position:

The patient is placed supine on the operating table and neck is positioned in extension so as to achieve optimum reduction. Intra-operative x-rays are obtained in the Antero_posterior and lateral planes.

Incision:

Longitudinal incision is made at the medial border of the sternomastoid muscle on the right side.The platysma is divided,and the fascia of the sternocleidomastoid is sharply incised along its medial border. Blunt dissection is used to expose the anterior surface of the spinal column at the midcervical level by opening natural planes medial to the carotid artery sheath and lateral to the trachea and esophagus.The fascia of the musculus longus colli is incised in the midline, and the muscle is elevated from the vertebra.Blunt dissection in the retropharyngeal space is used to open a tunnel in front of the vertebra to the C-2 level.

A K-wire is inserted through the incision up to the inferior edge of C-2, under Image, and impacted into the inferior edge of C-2. A K wire is advanced carefully controlled with biplane fluoroscopy from the inferior anterior edge of C-2 through the body of C-2 to the odontoid till its apex. A cannulated drill pit is then used over the wire. The drilled hole is then tapped. The screw, selected based on the measured depth, is placed and tightened firmly monitored fluoroscopically. One screw is biomechanically sufficient for fixation. The wound is checked for hemostasis,and closure completed in layers over a suction drain.

Post-operative care and follow up:

Post-operative collar for 6 weeks. Follow up visits at 2 weeks,2,6,12 months.Clinical and neurological assessment will be done and cervical X-rays will be ordered at each follow up visit.

Functional outcome will be evaluated by Association for the study of internal fixation(AO) neck pain and disability score postoperative and at 1 year follow up.

CT scan will be done for all patients at 1 year to ensure bony union.

ELIGIBILITY:
Inclusion Criteria:

_ All Type II odontoid fractures in adults .

Exclusion Criteria:

* Associated fracture body of C2 .
* Reverse type of odontoid fracture pattern.
* Pathological fractures or osteoporotic bone.
* Non-union.
* Short ,kyphotic neck and obese people.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases with type 2 odontoid fracture admitted to trauma unit assiut university hospital
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Association for the study of internal fixation(AO) neck disability index. | 1 year
  AO neck disability index is a questionnaire designed to give us information as to how neck pain has affected the ability to manage in everyday life. It consists of ten sections each of them descripes one of daily activity and graded from zero to five the higher the total score the more severity of disability. The sections are pain intensity, personal care , lifting, reading , headache, concentration, work, driving, sleaping, recreation . its developed by Vernon,H .& Mior,S . (1991)

SECONDARY OUTCOMES:
Assesment of bony union | 1year
  Measured by CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Fayez ahmed, Asyut, Nag Hamady, Egypt